CLINICAL TRIAL: NCT05225285
Title: Efficacy, Immunogenicity and Safety of Inactivated Vaccine (Coronavac) Against SARS-COV2 in Children and Adolescents - Curumim Project
Brief Title: Efficacy, Immunogenicity and Safety of Inactivated Vaccine (Coronavac) Against SARS-COV2 in Children and Adolescents
Acronym: Curumim
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Espirito Santo (Other)
Collaborators: Centro de Pesquisas René Rachou (Other Government); Butantan Institute (Other Government); Secretaria de Estado da Saúde do Espírito Santo - SESA (Unknown)
Responsible Party: Principal Investigator, Valéria Valim, Prof Dr, Federal University of Espirito Santo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FUES04
Record Dates: First submitted 2022-02-01; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: COVID-19
Keywords: covid-19; Vaccine; Children; Coronavac; Vero Cell
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 2 groups, in a 2:1 ratio, to receive the inactivated Coronavac/Butantan vaccine (VACC) and a group to receive the immunizing BNT162b2 (Pfizer) (BNTC). The VACC group will also be compared to a group of adults aged 18 to 49 who received Coronavac (ADU).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For blinding, the vaccine dose will be prepared by a pharmacist, who will be the only one who will know which immunizer will be administered. Vaccinators, participants and evaluators will not know which immunizer will be given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VACC (Experimental): This group will receive the inactivated Coronavac/Butantan vaccine.
  Interventions: Biological: Inactivated Coronavac/Butantan vaccine
- BNTC (Active Comparator): This group will receive the immunizing BNT162b2 (Pfizer).
  Interventions: Biological: BNT162b2 (Pfizer)
- ADU (Active Comparator): This group of adults participants will receive the inactivated Coronavac/Butantan vaccine.
  Interventions: Biological: Inactivated Coronavac/Butantan vaccine

INTERVENTIONS:
Biological: Inactivated Coronavac/Butantan vaccine — Inactivated Coronavac/Butantan vaccine in 2 doses of 0.5 ml, 4 weeks apart
  Arms: ADU; VACC
Biological: BNT162b2 (Pfizer) — BNT162b2 (Pfizer) vaccine in 2 doses of 0.1 ml or 0.30 ml (according to age group), 4 weeks apart
  Arms: BNTC

SUMMARY:
To evaluate the efficacy and safety of vaccinating children and adolescents, aged 3 to 17 years, with a two-dose schedule of the inactivated vaccine (Coronavac) against SARS-Cov-2.

DETAILED DESCRIPTION:
Nine hundred sixty (960) participants will be randomized into 2 groups, in a 2:1 ratio, to receive the inactivated Coronavac/Butantan vaccine (VACC, N=640) and a group to receive the immunizing BNT162b2 (Pfizer) (BNTC, N=320). The VACC group will also be compared to a group of adults aged 18 to 49 who received Coronavac (ADU, N=160). The main outcome will be the geometric title of neutralizing antibodies and the secondary outcomes will be the incidence of the number of cases confirmed by RT-PCR, the cellular immune response and frequency of adverse events. Outcomes will be evaluated before the first dose, and 28 and 90 days after the second dose, and followup after 6 and 12 months. The study hypothesis is that the cellular and humoral immune response of children and adolescents is not inferior to the age group 18 to 49 years, who received Coronavac and compared to children vaccinated with the immunizing BNT162b2 (Pfizer) and that the inactivated vaccine presents lower reactogenicity for the age group studied.

ELIGIBILITY:
Inclusion Criteria:

* Age between 3 and 17 years old (VACC and BNTC groups)
* Age between 18 and 49 years old (ADU group)

Exclusion Criteria:

* Pregnant teenagers;
* History of severe allergic reaction (anaphylaxis, urticaria or angioedema) to any previously administered vaccine;
* Have previously received a vaccine against COVID-19;
* Personal history of SARS-CoV-2-related Multisystem Inflammatory Syndrome (MIS-C);
* Immunosuppressed due to conditions such as inborn error of metabolism, HIV infection, neoplasia or use of immunosuppressive drugs (systemic corticosteroids for more than 14 days or another immunosuppressant).

Ages: 3 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1120 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-06-21 (Estimated); Study Completion 2023-03-21 (Estimated)

PRIMARY OUTCOMES:
Viral neutralization assay | 3 months
  Neutralizing antibody titers will be expressed by the ability of antibodies to neutralize up to 50% the number of plaques (PRNT50). Title > 1:50 will be considered positive.
Chemiluminescence serological assay for qualitative and quantitative determination of neutralizing antibodies against Spike protein (anti-SARS-Cov-2 anti-IgG-S) | 3 months
  Results are expressed in AU/mL and data interpretation will be as follows: <50 AU/mL = negative; ≥50 U/mL = positive.
Serological assay by chemiluminescence for qualitative and quantitative determination of specific IgG antibodies against the nucleocapsid protein of SARS-Cov-2 | 3 months
  Results will be expressed as fluorescence intensity or pg/mL. The cutoff is 1.4 and <1.4 = negative; ≥1.4 = positive.
Dosage of systemic soluble factors | 12 months
  Chemokines, cytokines and growth factors - biomarkers of humoral and cellular response. Results will be expressed in pg/mL.
Antigen-specific stimulation of peripheral blood mononuclear cells in vitro | 2 months
  The results will be expressed as a positive percentage frequency for a given cell phenotype.
T lymphocytes | 12 months
  The results will be expressed as a positive percentage frequency for a given cell phenotype.
B lymphocytes | 12 months
  The results will be expressed as a positive percentage frequency for a given cell phenotype.
intracytoplasmic cytokines | 12 months
  The results will be expressed as a positive percentage frequency for a given cell phenotype.

SECONDARY OUTCOMES:
RT-PCR confirmed cases | 6 months
  Cases confirmed by RT-PCR, whose signs/symptoms have started 15 days after the second dose of vaccine, over 6 months after receiving the vaccine.
Adverse events | 6 months
  Surveillance of adverse post-vaccine events (PVAE) and adverse events of special interest (EAIE) will be carried out.

CONTACTS AND LOCATIONS:
Locations (1):
- Valéria Valim, Vitória, Espírito Santo, Brazil

IPD SHARING:
Plan to Share IPD: No